CLINICAL TRIAL: NCT05425290
Title: Emotion Regulation Training to Reduce Cardiovascular Disease Risk Among Depressed Young Adults in Southern Mississippi: A Single-Session Design
Brief Title: Emotion Regulation Training to Reduce Cardiovascular Disease Risk Among Depressed Young Adults in Southern Mississippi
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Mississippi (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: USMississippi
Record Dates: First submitted 2022-02-20; First posted 2022-06-21 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Major Depressive Disorder; Cardiovascular Diseases; Inflammation; Blood Pressure; Heart Rate Variability
MeSH Terms: conditions — Depressive Disorder, Major; Cardiovascular Diseases; Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Arm (Experimental)
  Interventions: Behavioral: Single-session emotion regulation training

INTERVENTIONS:
Behavioral: Single-session emotion regulation training — The single-session emotion regulation skills training will blend psychotherapeutic approaches that emphasize effective ER. First, participants will be taught to adopt a detached (i.e., 'distanced') and nonjudgmental attitude towards an emotional situation. Detachment, or 'distancing' as it will be introduced to participants, will be taught by examining the situation with objectivity or putting spatial or temporal distance between the current moment and the situation. Second, research participants will be taught reframing. Specifically, they will be introduced to the relationship between thoughts and emotions and how to find interpretations that are less upsetting in order to be more effective when upset. Participants will identify elements of a situation that they did not pay attention to or information that was missing, and to reframe their thoughts based on the full picture. The emotion regulation training is expected to take approximately 30-45 minutes.

SUMMARY:
The proposed study will investigate the utility of a single-session emotion regulation training to reduce CVD risk among young adults diagnosed with MDD living in Southern MS. Using an single-arm, non-randomized design, young adults aged 18-29 will undergo a single-session emotion regulation skills training. Before and immediately after the skills training session, participants will supply several biological metrics tied to CVD risk: resting HRV, inflammation (measured via c-reactive protein [CRP]), and blood pressure. Participants will provide the same biological metrics at a one-week follow-up visit to assess short-term sustained gains following the single-session intervention and complete a 7-day ecological momentary assessment (EMA) of their daily emotion regulation skills use and depressive symptoms between these two visits.

DETAILED DESCRIPTION:
Cardiovascular disease (CVD) is a leading cause of death in Mississippi, accounting for over a third of deaths within the state. Mississippians face numerous health disparities that enhance disease risk throughout our community. In addition to behavioral factors, several notable biological markers enhance risk for CVD including low resting heart rate variability (HRV), high blood pressure, and inflammation. In Mississippi, an estimated 20.9% of adults meet criteria for depression. Adults experiencing depressive disorders experience high rates of emotion dysregulation, and psychological interventions that include emotion regulation training components are highly efficacious in reducing psychological and physical symptoms associated with depression. Depression, particularly major depressive disorder, is routinely linked with enhanced CVD risk. Understanding and intervening on the relationship between CVD risk factors and depression in young adulthood offers potential to prevent exacerbation of risk later in life. This pilot study will investigate the utility of a single-session emotion regulation training to reduce CVD risk among young adults living in Southern Mississippi who are diagnosed with major depressive disorder (MDD). The study aims are to: 1) examine whether the single-session emotion regulation training promotes changes in biological risk factors for cardiovascular disease immediately following the training and at a 1-week follow-up visit; 2) to assess whether the single-session emotion regulation training reduces depressive symptoms among research subjects; and 3) to test whether use of emotion regulation skills learned during the training in the week following the intervention session promotes greater changes in cardiovascular disease risk factors. Using a lab-based experimental intervention design, young adults will undergo a single-session emotion regulation skills training. Before and after the skills training session, research subjects will supply several physiological metrics tied to CVD risk: resting HRV, c-reactive protein (CRP) levels, and blood pressure. Subjects will provide the same biological metrics at a one-week follow-up visit to assess short-term sustained gains following the single-session intervention. Results from this study offer potential to reduce emotion regulation difficulties associated with major depression, reduce CVD risk factors among young adults in Mississippi, and advance our knowledge of how psychological interventions can improve both psychological and physical risk factors for chronic health conditions among young adults, potentially buffering depression's long-term health impact.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women ages 18-29
2. Able to speak and read English
3. Outpatient at the time of participation
4. Able to provide informed consent
5. Stable medications for 30 days or more
6. Appropriate diagnoses:

   * Meets diagnostic criteria for current major depressive disorder

Exclusion Criteria:

1. Not fluent in English
2. Not able to provide informed consent
3. Active suicidal ideation
4. Presence of autoimmune and/or inflammatory diseases (e.g., rheumatoid arthritis, ulcerative colitis)
5. Ongoing use of steroids (if use of steroids is temporary, individuals are eligible to participate 30 days after termination)
6. Medication change in the past 30 days (individuals are eligible to participate 30 days after a medication change and may take advantage of delayed scheduling)
7. Meets diagnostic criteria for a schizophrenia-spectrum disorder, substance use disorder, and/or bipolar disorder
8. Presence of a cardiovascular disease (e.g., hypertension) or prescribed cardiovascular medications (e.g., beta blockers, blood pressure medication)

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2022-08-25 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Diastolic Blood Pressure | Change from prior to the single-session emotion regulation training to immediately after and 1-week after
  Diastolic blood pressure will be measured prior to the training, immediately afterwards, and during the 1-week follow-up visit
Change in Systolic Blood Pressure | Change from prior to the single-session emotion regulation training to immediately after and 1-week after
  Systolic blood pressure will be measured prior to the training, immediately afterwards, and during the 1-week follow-up visit
Change in Resting Heart Rate Variability (HRV) | Change from prior to the single-session emotion regulation training to immediately after and 1-week after
  Resting heart rate variability (HRV) will be measured prior to the training, immediately afterwards, and during the 1-week follow-up visit
Change in C-reactive protein (CRP) | Change from prior to the single-session emotion regulation training to immediately after and 1-week after
  C-reactive protein (CRP) will be measured prior to the training, immediately afterwards, and during the 1-week follow-up visit
Change in Center for Epidemiological Studies - Depression Scale (CESD) | Change from prior to the single-session emotion regulation training to immediately after and 1-week after
  Depressive symptoms will be assessed using the CESD prior to the training, immediately afterwards, and at the 1-week follow-up visit. Depressive symptoms will also be assessed during the EMA assessment period.

SECONDARY OUTCOMES:
Change in Emotion Regulation Questionnaire, Reappraisal subscale (ERQ-R) | Change from prior to the single-session emotion regulation training to immediately after and 1-week after
  Reappraisal Skills will be measured by the ERQ-R and assessed prior to the training, immediately afterwards, and at the 1-week follow-up visit. Reappraisal skills will also be assessed during the EMA assessment period.
Change in Experiences Questionnaire - Decentering (EQ-D) | Change from prior to the single-session emotion regulation training to immediately after and 1-week after
  Decentering skills, measured by the EQ-D, will be assessed prior to the training, immediately afterwards, and at the 1-week follow-up visit. Decentering skills will also be assessed during the EMA assessment period.
Change in Difficulties with Emotion Regulation Scale (DERS) | Change from prior to the single-session emotion regulation training to immediately after and 1-week after
  Emotion Dysregulation, measured by the DERS, will be assessed prior to the training, immediately after, and at the 1-week follow-up visit.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Southern Mississippi, Hattiesburg, Mississippi, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data will be available upon reasonable request.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code